CLINICAL TRIAL: NCT00065078
Title: Effectiveness of Nurse Home Contraceptive Dispensing
Brief Title: Providing Birth Control Through Home Health Visits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD042423 (NIH)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Pregnancy
Keywords: Home-visits; Community nurse; Unintended pregnancy

INTERVENTIONS:
Procedure: Home dispensing of contraception

SUMMARY:
This study will evaluate a program that provides birth control to low income and minority women through home visits by a community health nurse. The goal of the program is to reduce unwanted pregnancies.

DETAILED DESCRIPTION:
Unintended pregnancy is associated with significant public health problems, including inadequate prenatal care, low birth weight infants, infant mortality, and maternal morbidity and mortality. Children born as a result of unplanned pregnancies are at greater risk for poor outcomes such as poor mental health and developmental disabilities. This research project will determine whether providing contraception in the home can reduce the incidence of unintended pregnancy in low income and minority women. The project will also determine whether delaying a pelvic exam encourages or discourages the utilization of clinic-based preventive services to screen for sexually transmitted diseases (STDs) and cervical cancer.

Participants will be randomized to either an experimental group or a comparison group. Each participant will receive family planning counseling during a home visit by a community health nurse. Participants in the experimental group will be offered a three-month supply of oral contraceptives or a depo-provera shot; both forms of contraceptives will be delivered during home visits. Each participant will complete a survey during the initial visit and during a 1-year follow-up. The study will last approximately three years.

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing age
* Not pregnant
* Interested in delaying pregnancy using oral contraceptives or a depo-provera shot
* Had sex in the last month or are planning to have sex in the next month
* Have not used contraception during every sexual encounter within 3 months prior to study entry

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2003-06; Study Completion 2005-07

PRIMARY OUTCOMES:
Pregnancy

SECONDARY OUTCOMES:
Sexually Transmitted Disease Screening

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Melnick, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Clackamas County Public Health Division, Oregon City, Oregon, United States